CLINICAL TRIAL: NCT05733910
Title: Simultaneous Integrated Boost (SIB) Planning Approach in Carbon Ion Radiotherapy for Head and Neck Adenoid Cystic Carcinoma
Brief Title: Simultaneous Integrated Boost in Carbon Ion Radiotherapy for Head and Neck Adenoid Cystic Carcinoma
Acronym: SIBACIRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CNAO 46 2022C
Record Dates: First submitted 2023-01-24; First posted 2023-02-17 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma, Adenoid Cystic; Head and Neck Cancer
Keywords: adenoid cystic carcinoma; hadrontherapy; carbon ion radiation therapy CIRT; head and neck cancer; SIB
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: The patients will be prospectively enrolled and treated at the sponsor's premises. Only one group of subjects will enter the phase II trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- carbon ion radiotherapy (Experimental): simultaneous integrated boost with carbon ion radiotherapy
  Interventions: Radiation: simultaneous integrated boost of carbon ions radiation therapy

INTERVENTIONS:
Radiation: simultaneous integrated boost of carbon ions radiation therapy — CIRT Treatment will be delivered in 16 fractions, 4 fractions per week. Treatment plans will be calculated with a Simultaneous Integrated Boost Approach (SIB).
  The HR-CTV will receive a total dose of 65.6 GyRBE (4.1 GyRBE/fraction). The LR-CTV will simultaneously receive a total dose of 54.4 GyRBE (3.4 GyRBE/fraction) or 48 GyRBE (3 GyRBE/fraction) at discretion of Radiation Oncologist depending on the prognostic factors (54.4 GyRBE in case of macroscopical perineural invasion or positive margin along the nerve, 48.0 Gy(RBE) in case of elective perineural irradiation or microscopic focal intratumor perineural invasion).
  Other Names: CIRT

SUMMARY:
The investigators aim at investigating in a prospective clinical trial whether using a Simoultaneous Integrated Boost of carbon ions treatment planning approach, improving the tumor dose conformation while lowering the unintended dose to the low-risk volume, can significantly reduce the probability of toxicity without affecting Local Control.

DETAILED DESCRIPTION:
In photon radiotherapy, Simultaneous integrated boost (SIB)-intensity-modulated radiation therapy (IMRT) with slight hypofractionation in the HR-CTV is the current standard of care, being previously largely adopted in clinical practice and within several prospective clinical trials, with similar results in terms of toxicity and oncologic outcome.

Up to now, a simultaneous integrated boost (SIB) approach has not been fully exploited in CIRT so far. The expected benefit of a SIB planning approach in carbon ion treatment is the reduction of toxicity with respect to the sequential (SEQ) approach currently used in CNAO clinical practice, while maintaining the same local control rate. This benefit depends on the potentiality of SIB to better spare normal tissues, further enhancing the intrinsic favourable physical and radiobiological characteristics of the carbon ions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven primary head and neck ACC;
* Unresectable stage or residual macroscopic disease after surgery or multiple microscopic margins after surgery;
* Patient with resectable tumor but refusing surgery
* cN0/pN0 - cN1/pN1 patients (only ipsilateral neck levels I and II)
* Absence of distant metastases or oligometastatic status (patients with ≤ 3 metastatic lung or bone lesions, excluding other sites;
* No previous radiotherapy in head and neck region;
* Karnofsky Performance Status ≥ 70;
* Age ≥ 18 years;
* Written informed consent
* Patients' ability to understand the characteristics and consequences of the clinical trial.

Exclusion Criteria:

* Local conditions contraindicating CIRT (e.g., active infection or previous history of recurrent infections in or close to the tumor site; intratumoral necrosis in strict proximity of vessels; pre-existing skin, bone or soft tissue fistula; extended mucosal involvement by the tumor; previous surgery with flap reconstruction);
* Tumour site in nasopharynx, pharynx and tongue base (where an exclusive CIRT treatment could be at high risk of toxicity);
* Tumor disease involving ≥ 50% of the palate with consequent high risks of serious anatomical damage in case of significant and rapid disease response to CIRT
* Nodal involvement > cN1/pN1 or cN1/pN1 outside ipsilateral levels I and II
* Tumor surrounding carotid artery > 180° or infiltrating the vessels
* itanium surgical implants or metal prostheses or any other condition that prevents adequate imaging to identify the target volume and may determine uncertainties in CIRT dose distribution during treatment planning
* Presence of any comorbidity deemed to impact on treatment toxicity;
* Psychic or other disorders that may prevent informed consent
* Active autoimmune disease (e.g. systemic lupus erythematosus, systemic sclerosis, rheumatoid arthritis)
* Contraindication to MRI
* Pregnancy or breastfeeding in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
acute and sub acute toxicity as assessed by CTACE 5.0 | 90 and 180 days after radiation treatment
  Acute and subacute toxicity will be assessed with clinical evaluation within 180 days after the end of treatment and graded using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
local control assessed through head and neck MRI | from last day of radiation treatment up to 12 months until disease progression or death or last follow up up to 5 years
  LC is expected to be the same as in the sequential traditional approach
toxicity evaluation | toxicity assessed at 90, 120, 180 days
  various toxicity endpoints will be aggregated and analysed to build predictive factors to build multivariate predictive models

CONTACTS AND LOCATIONS:
Overall Officials: Sara Ronchi, MD, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Pavia, Italy